CLINICAL TRIAL: NCT03789669
Title: A Prospective, Multi-Center Evaluation of Corneal Flap Creation Using Cheetah Femtosecond Laser System and Cheetah Patient Interface
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Surgical Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHTA-103-FLAP
Record Dates: First submitted 2018-12-27; First posted 2018-12-28 (Actual); Results first posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Refractive Error
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Investigational/Control (Active Comparator): Both eyes of each subject will be treated. The investigators will use the investigational Cheetah femtosecond laser and Cheetah PI on one eye, and commercial iFS femtosecond laser and PI on the other eye to create a LASIK flap on subjects' corneas. Flap parameters (such as flap depth, flap diameter, and hinge angle) should be the same for both eyes. The eye to receive Cheetah flap will be randomized (ratio of 1:1 for right eye and left eye).
  Subjects will undergo refractive correction via corneal ablation on both eyes using a commercial excimer laser for vision correction (same excimer laser system will be used on both eyes).
  Interventions: Device: IntraLase iFS femtosecond laser and patient interface
- Control/Investigational (Active Comparator): Both eyes of each subject will be treated. The investigators will use the commercial Cheetah femtosecond laser and Cheetah two piece PI on one eye, and commercial Cheetah femtosecond laser and investigational Cheetah to create a LASIK flap on subjects' corneas. Flap parameters (such as flap depth, flap diameter, and hinge angle) should be the same for both eyes. The eye to receive Cheetah flap will be randomized (ratio of 1:1 for right eye and left eye).
  Subjects will undergo refractive correction via corneal ablation on both eyes using a commercial excimer laser for vision correction (same excimer laser system will be used on both eyes).
  Interventions: Device: Cheetah femtosecond laser and cheetah patient interface

INTERVENTIONS:
Device: IntraLase iFS femtosecond laser and patient interface — Commercial ophthalmic laser surgical system
  Arms: Investigational/Control
Device: Cheetah femtosecond laser and cheetah patient interface — Ophthalmic laser surgical system
  Arms: Control/Investigational

SUMMARY:
The study is a prospective, open-label, comparative study design that was chosen for the purpose of optimizing the Cheetah settings, and evaluating the Cheetah system quality of LASIK flap.

DETAILED DESCRIPTION:
This study is a 3-month, prospective, multicenter, open-label, comparative, randomized (1:1 ratio for right and left eyes) study.

The study will be conducted at up to 5 sites and up to 300 treated subjects to achieve minimum 40 eyes with optimized settings and additional eye data for further device experience.

Both eyes of each subject will be treated. The investigator will use the Cheetah femtosecond laser, with the following possible procedures performed:

A comparison of commercial iFS femtosecond laser and PI in one eye and the Cheetah femtosecond laser (with the two piece PI) on the other eye. The eye treated with the Cheetah femtosecond laser will be the study eye and the eye treated with the commercial iFS femtosecond laser will be the control eye.

All procedures will be performed to create a LASIK flap on subjects' corneas. Flap parameters (such as flap depth, flap diameter, and hinge angle) should be the same for both eyes. The study eye will be randomized (ratio of 1:1 for right eye and left eye).

Subjects will undergo refractive correction via corneal ablation on both eyes using a commercial excimer laser for vision correction (same excimer laser system shall be used on both eyes).

Over the course of the study, minor prototype device settings/improvements (with no safety implications and without compromising the clinical validity of the study) may be performed to optimize the quality of flap.

ELIGIBILITY:
INCLUSION CRITERIA

To be considered for enrollment of the study, subject must:

* Sign an informed consent and HIPAA authorization
* Be at least 18 years of age at the time of study exam
* Have refractive error and be eligible for commercial LASIK treatment
* Be available for all scheduled follow-up visits (see below)

EXCLUSION CRITERIA

Subject will not be eligible to take part of the study if subject, use or have:

* Known to be pregnant, breastfeeding or intend to become pregnant during the study.
* Recent ocular (eye) trauma or eye surgery
* A history of or active ophthalmic (eye) disease or abnormality
* Ocular hypertension (high eye pressure) with IOP (eye pressure) greater than 21 mmHg, glaucoma suspect, or are taking medications for these conditions
* A history or current diagnosis of any of the following medical conditions that could affect wound healing: collagen vascular disease, autoimmune disease, immunodeficiency disease, ocular herpes; endocrine disorders including, but not limited to unstable thyroid disorders and diabetes, lupus, and rheumatoid arthritis.
* Cardiac pacemaker, implanted defibrillator or other implanted electronic device
* Taking systemic or inhaled medications that may affect wound healing
* Known sensitivity or inappropriate responsiveness to any of the medications used in the study
* Desire for monovision correction
* Participating in any other clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Surgical Vision Clinical Trials, Study Director — Johnson & Johnson Surgical Vision
Locations (3):
- India (2):
  - Narayana Nethralaya Eye Hospital, RajajiNagar, Bangalore
  - Center For Sight, Safdarjung Enclave, New Delhi
- Tan Tock Seng Hospital PTE. LTD., Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a paired-eye study design in which for each subject, one eye is treated with ELITA and the fellow eye is treated with iFS. For the primary endpoints, a relative scale of 1-5 was used to compare the performance of the ELITA treated eye vs iFS treated eye. The primary endpoint evaluations require both eyes to be treated; thus, 3 unilaterally treated subjects were excluded from the analysis. There is only one arm for primary endpoint evaluation; and two arms for other analyses.
Pre-assignment Details: A total of 200 subjects were enrolled in the study. 45 subjects were consented but not treated in the study. 3 subjects were one-eye treated with ELITA; and 197 subjects were treated bilateral (one eye treated with ELITA, one eye treated with controlled system iFS). 3 unilaterally treated subjects were excluded from the analysis. A score of 4 or 5: study eye was better than the control eye. A score of 3: equal performance. A score of 1 or 2: study eye was worse than the control eye.
Units Other Than Participants: Eyes
Groups:
- Unilateral: ELITA - One Eye Treated with ELITA, Fellow Eye Not Treated
- Bilateral: One eye treated with ELITA, fellow eye treated with iFS
Period: Overall Study
Arm/Group | Unilateral | Bilateral
Started | 3; 3 Eyes | 197; 394 Eyes
Completed | 0; 0 Eyes | 197; 394 Eyes
Not Completed | 3; 3 Eyes | 0; 0 Eyes

BASELINE CHARACTERISTICS:
Population: 3 unilaterally treated subjects were excluded in analysis as they were not applicable.
Units Other Than Participants: Eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | Unilateral | Bilateral | Total
Number analyzed (Participants) | 3 | 197 | 200
Number analyzed (Eyes) | 3 | 394 | 397
Age, Customized [Count of Participants; unit: Participants]
  >=50 years old | 0 | 0 | 0
  40-49 years old | 0 | 3 | 3
  30-39 years old | 1 | 53 | 54
  <30 years old | 2 | 141 | 143
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 95 | 97
  Male | 1 | 102 | 103
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 197 | 200
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 197 | 200
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Stromal Bed Surface Quality
Description: Surface quality will be graded on a scale of 1-5 relative to Intralase iFS flap. Number of Participants with Stromal Bed Surface Quality scale of 3 or higher.
Time Frame: At the Operative visit, one time visit
Population: 3 unilaterally treated subjects were excluded from the analysis. There is only one arm analyzed for primary outcome measure. The primary endpoint evaluations require both eyes to be treated.
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Unilateral | Bilateral
Number analyzed (Participants) | 0 | 197
Number analyzed (Eyes) | 0 | 394
Eyes | 0 | 175

2. Other Pre Specified Outcome: Flap Thickness
Description: The central flap thickness is measured per each eye, compared from ELITA vs. iFS performances.
Time Frame: 3 months
Population: This Outcome Measure has different Group from the Outcome Measure 1, Test Group with one eye with ELITA and Control Group, the fellow eye with the iFS. At 3-month visit, there were only 132 participants in the analysis. These data were not collected from participants in the Unilateral group.
Measure: Mean (Standard Deviation); unit: microMeter
Units Other Than Participants: Eyes
Groups:
- Test: One Eye Treated with ELITA
- Control: Fellow Eye Treated with iFS
Arm/Group | Test | Control
Number analyzed (Participants) | 132 | 132
Number analyzed (Eyes) | 132 | 132
microMeter | 109.32 (6.55) | 109.77 (6.53)

ADVERSE EVENTS:
Time Frame: During the course of the study until termination (3 months)
Description: Adverse events were not monitored or assessed at the eye level and cannot be attributed to a specific intervention. AEs were monitored/ assessed at the participant level.
  3 unilaterally treated subjects - 3 eyes in total from 3 participants; 197 bilaterally treated subjects - 394 eyes in total from 197 participants.
Groups:
- Unilateral: One eye treated with ELITA only, Fellow Eye Not Treated
Arm/Group | Unilateral | Bilateral
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/197
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/197
Other Adverse Events (participants affected / at risk) | 3/3 | 2/197
OTHER ADVERSE EVENTS (reported when occurring in more than 0.15% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Unilateral (N=3) | Bilateral (N=197)
Miscreated Flap (Surgical and medical procedures) | 1 | 0
Epithelium in the interface with a loss of 2 or more lines of BSCVA (>10 ETDRS letters) (Surgical and medical procedures) | 0 | 1
Other (Surgical and medical procedures) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2023-05-05): https://cdn.clinicaltrials.gov/large-docs/69/NCT03789669/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-06): https://cdn.clinicaltrials.gov/large-docs/69/NCT03789669/SAP_001.pdf